CLINICAL TRIAL: NCT03038282
Title: Effects of Chromium on Insulin Resistance in Alzheimer Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Metabolic Therapy Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01TCR012617
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — chromous chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chromium Chloride (Experimental): Participants transdermal chromium chloride 50 to 600 mcg/day.
  Interventions: Dietary Supplement: Chromium Chloride
- Individual Exercise (Experimental): Exercise 150 minutes per week (over 3 to 5 days) for 12 weeks.
  Interventions: Other: Individual Exercise
- Control Group (No Intervention): Participants or participant's caregiver will be provided educational materials on starting an exercise program and instructions for the application of transdermal chromium chloride, but will receive no formal support for their exercise program.

INTERVENTIONS:
Dietary Supplement: Chromium Chloride — Transdermal chromium chloride 50 to 600 mcg/day.
  Arms: Chromium Chloride
Other: Individual Exercise — Participants will engage in 150 minutes of exercise over 3-5 days per week for 12 weeks
  Arms: Individual Exercise

SUMMARY:
The effect of Chromium to improve glucose levels in Alzheimer Disease (AD) is controversial. The hypothesis of the study is to evaluate the effect of supplementing the AD individuals with Chromium combined with exercise and assessing the effect of the supplementation on glucose metabolism.

DETAILED DESCRIPTION:
Chromium is an essential nutrient required for optimal insulin activity and normal carbohydrate and lipid metabolism. Beyond its nutritional effects, dietary supplement of chromium causes beneficial outcomes against several diseases, in particular diabetes-associated complications such as Alzheimer Disease. Common forms include chromium chloride, chromium nicotinate, and chromium picolinate.

The argument for chromium supplementation relies on evidence from case reports of resolution of diabetic symptoms refractory to insulin via chromium added to total parenteral nutrition, and experiments in which animals deficient in chromium exhibited impaired glucose metabolism.

Chromium may influence glucose metabolism by increasing the number of insulin receptors or by binding insulin to receptors. The US Food and Drug Administration concludes that, based on recent studies, chromium picolinate may reduce the risk of insulin resistance and therefore may reduce the risk of type 2 diabetes.

A number of systematic reviews and meta-analyses have been conducted to determine the effect of chromium on glycemic control, although large, quality trials are limited. The majority of studies have found no effect on measured outcomes, with a few studies contributing to the positive observed effects. Variations of preparations used in the trials and study conditions make generalization of the results difficult.

In order to provide a comprehensive clinical evaluation of the effects of Chromium in AD patients, we will conduct a double-blinded and placebo-controlled trial in subjects with AD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Alzheimer's disease.
* Exhibiting an onset and progression of cognitive dysfunction during at least 3 months prior to the screening period.

Exclusion Criteria:

* Patients with neurodegenerative diseases other than Alzheimer's disease.
* Patients with cognitive dysfunction due to cerebral damage resulting from a lack of oxygen, a brain injury, etc.
* Patients with clinically significant cardiovascular disease.
* Patients with history of clinically-evident stroke.
* Patients with history of cancer in the last 5 years.
* Patients with clinically-significant systemic illness that may affect safety or completion of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance | Change from Baseline to 12 weeks
  Insulin action will be determined by insulin clamp and OGTT using deuterated glucose both before and after treatment.

SECONDARY OUTCOMES:
Change in chronic refractory mood disorders | Change from Baseline to 12 weeks
  To be measured using confirmatory factor analysis (CFA). CFA aggregates scores from across multiple subtests.

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Haley, PhD, Principal Investigator — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: Undecided
Sharing data will be available upon written request.